CLINICAL TRIAL: NCT04755088
Title: A Phase 1 Study To Assess The Effect Of Moderate Renal Impairment On The Pharmacokinetics Of Surufatinib
Brief Title: Surufatinib Renal Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-012-00US3
Record Dates: First submitted 2021-02-04; First posted 2021-02-15 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Subjects with Normal Renal Function: All patients to receive study drug (Surufatinib 300mg) on Day 1
  Interventions: Drug: Surufatinib
- Cohort 2 (Experimental): Subjects with Moderate Renal Impairment: All patients to receive study drug (Surufatinib 300mg) on Day 1
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Subjects to receive Surufatinib 300mg on Day 1
  Other Names: HMPL-012
  Arms: Cohort 1
Drug: Surufatinib — Subjects to receive Surufatinib 300mg on Day 1
  Other Names: HMPL-012
  Arms: Cohort 2

SUMMARY:
An open-label, multicenter, single-dose, single-period, sequential study to assess the effect of moderate renal impairment on the pharmacokinetics of surufatinib.

DETAILED DESCRIPTION:
An open-label, multicenter, single-dose, single-period, sequential study with the primary objective of assessing the effect of moderate renal impairment on the PK of surufatinib following administration of 300mg single oral dose. The secondary objective is to evaluate the safety in subjects with moderate renal impairment and subjects with normal renal function following a single oral dose of 300mg surufatinib.

Approximately 16 subjects will be enrolled

ELIGIBILITY:
Inclusion Criteria:

All subjects

* The subject is male or female between the ages of 18 and 79 years old (inclusive).
* The subject has a BMI >18 and ≤40 kg/m2 and body weight not <50 kg at screening.
* The subject is a non-smoker or light smoker who smokes no more than 10 cigarettes, 2 cigars, 2 pipes, or other nicotine equivalents (eg, vape, snuff, gum) of tobacco per day; willing to limit smoking during the treatment period to 4 cigarettes or 1 cigar per day.
* Females must be of non-childbearing potential or surgically sterile
* Males who have not had a successful vasectomy and are partners of women of childbearing potential must use, or their partners must use, a medically acceptable method of contraception starting for at least 1 menstrual cycle prior to and throughout the entire study treatment period and for 2 weeks after the last dose of study drug. Those with partners using hormonal contraceptives must also use an additional approved method of contraception, such as a condom with spermicide. Males who have had a successful vasectomy (confirmed azoospermia; documentation needed) require no additional contraception. No sperm donation is allowed during the study treatment period and for 90 days after study drug discontinuation. Males must confirm that female partners of childbearing potential agree to use medically accepted contraception methods.

Subjects with Moderate Renal Impairment

* The subject must have eGFR of 30-59 mL/min/1.73 m^2 as calculated by MDRD.
* The subject must have no clinically significant change in disease status within the last 30 days before screening.
* If diabetic, the subject must have the disease controlled
* The subject must have blood pressure between 90 and 160 mm Hg systolic, inclusive, and not higher than 100 mm Hg diastolic.

Subjects with Normal Renal Function

* The subject must be without renal disease and have normal renal function (eGFR ≥90 mL/min/1.73 m2 based on the MDRD equation) at screening and check-in. Clinical laboratory test results must be within the normal laboratory reference ranges for serum urea, serum protein, and serum albumin.
* The subject must be without renal disease and have normal renal function
* The subject must be in good health
* The subject must have blood pressure between 95 and 150 mm Hg systolic, inclusive, and no higher than 90 mm Hg diastolic

Exclusion Criteria:

All Subjects

* The subject has evidence of clinically significant cardiovascular, hepatic, GI, respiratory, endocrine, hematological, neurological, or psychiatric disease or abnormalities.
* The subject has a clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to the first dose.
* The subject has a clinically significant ECG abnormality
* The subject has been diagnosed with acquired immune deficiency syndrome (AIDS), or tests positive for human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
* The subject has participated in a clinical study of another drug before dosing, and the time since the last use of other study drug is less than 5 times the half-life or 4 weeks before Day 1, whichever is longer, or is currently enrolled in another clinical study.
* The subject has consumed grapefruit, starfruit, Seville oranges, or their products within 7 days prior to the first dose.
* The subject has consumed herbal preparations/medications, including, but not limited to, kava, ephedra (ma huang), Ginkgo biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng, within 7 days prior to the first dose.
* The subject has received blood or blood products within 8 weeks, or donated blood or blood products within 8 weeks prior to the first dose, or donated double red cells within 16 weeks prior to the first dose.
* The subject has experienced a weight loss or gain of >10% within 4 weeks prior to the first dose.
* The subject has used any drug that is a strong inhibitor or inducer (including St. John's wort) of CYP3A or P-gp within 2 weeks prior to first dose or will require use during study treatment period.
* The subject is allergic to the study drug or to any of its excipients.
* Female subjects who are pregnant or planning to become pregnant, lactating, or breastfeeding.
* The subject has used a proton pump inhibitor (PPI) within 4 days prior to the first dose or a histamine 2 (H2) receptor antagonist (H2 blocker) within 2 days prior to the first dose.

Subjects with Moderate Renal Impairment

* The subject has clinically significant vital sign abnormalities at screening or baseline.
* The subject has a history of drug or alcohol misuse within 6 months prior to screening or a positive drug test at screening or Day -1.
* The subject has clinically significant physical, laboratory, or ECG findings
* The subject has any history of renal transplant.
* The subject has any known significant bleeding diathesis (eg, history of recent bleeding from esophageal varices) that could preclude multiple venipuncture or deep intramuscular injections.
* The subject has acute or exacerbating renal disease, fluctuating or rapidly deteriorating renal function as indicated by widely varying or worsening of clinical and/or laboratory signs of renal impairment within 2 weeks of first dose.

Subjects with Normal Renal Function

* The subject has evidence of clinically significant renal disease or abnormalities.
* The subject has evidence of a clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations at screening or baseline.
* The subject has a history of drug or alcohol misuse within 6 months prior to screening or a positive drug test at screening or Day -1.
* The subject has used any prescription or nonprescription drugs, including over-the-counter (OTC) medications or vitamins, within 2 weeks prior to the first dose.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2021-08-21 (Actual)

PRIMARY OUTCOMES:
AUC0-t | From Day 1 to Day 5 for Normal Renal Function; From Day 1 to Day 6 for Moderate Renal Impairment
  Area under the plasma concentration time curve from time 0 to the last measurable concentration
AUC0-inf | From Day 1 to Day 6
  Area under the plasma concentration time curve from time 0 to infinity (if data permit)
Cmax | From Day 1 to Day 6
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events as assessed by NCI CTCAE v5.0 | From Day 1 to Day 6
  To evaluate the safety of a single dose of 250 mg surufatinib administered in healthy subjects with normal renal function and subjects with moderate renal impairment.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orange County Research Center, Tustin, California
  - Orlando Clinical Research Center, Inc., Orlando, Florida